CLINICAL TRIAL: NCT03948113
Title: Outcome of Autosomal Dominant Polycystic Kidney Disease Patients on Peritoneal Dialysis: a National Retrospective Study Based on Two French Registries (the French Language Peritoneal Dialysis Registry and the French Renal Epidemiology and Information Network).
Acronym: ADPKDPD
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: 2018Ao005
Record Dates: First submitted 2019-05-10; First posted 2019-05-13 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Polycystic Kidney Diseases
MeSH Terms: conditions — Polycystic Kidney Diseases | interventions — Dialysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Dialysis

SUMMARY:
Pathological features of Autosomal Dominant Polycystic Kidney disease (ADPKD) include enlarged kidney volume, a higher frequency of digestive diverticulitis and abdominal wall hernias. Therefore, many nephrologists have concerns about the use of peritoneal dialysis (PD) in ADPKD patients. We aimed to analyze survival and technique failure in ADPKD patients treated with PD.

DETAILED DESCRIPTION:
Pathological features of Autosomal Dominant Polycystic Kidney disease (ADPKD) include enlarged kidney volume, a higher frequency of digestive diverticulitis and abdominal wall hernias. Therefore, many nephrologists have concerns about the use of peritoneal dialysis (PD) in ADPKD patients. We aimed to analyze survival and technique failure in ADPKD patients treated with PD. We conducted two retrospective studies on patients starting dialysis between 2000 and 2010, and based on two French registries: The French Renal Epidemiology and Information Network (REIN) and The French Language Peritoneal Dialysis Registry (RDPLF).

ELIGIBILITY:
Iinclusion criteria :

* Patients starting dialysis
* Patients included from the French Renal Epidemiology and Information Network (REIN) and The French Language Peritoneal Dialysis Registry (RDPLF) exclusion criteria
* patients without diagnosis of nephropathy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients starting dialysis and included from the French Renal Epidemiology and Information Network (REIN) and The French Language Peritoneal Dialysis Registry (RDPLF)
Sampling Method: Non-Probability Sample
Enrollment: 17350 (Actual)
Dates: Start 2000-02 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Overall survival | 15 years
  the time from the start of dialysis to death

SECONDARY OUTCOMES:
technique survival | 15 years
  the time from the start of dialysis to change of dialysis technique (death and transplantation were considered as competing risk)

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sigogne M, Kanagaratnam L, Dupont V, Couchoud C, Verger C, Maheut H, Hazzan M, Halimi JM, Barbe C, Canivet E, Petrache A, Drame M, Rieu P, Toure F. Outcome of autosomal dominant polycystic kidney disease patients on peritoneal dialysis: a national retrospective study based on two French registries (the French Language Peritoneal Dialysis Registry and the French Renal Epidemiology and Information Network). Nephrol Dial Transplant. 2018 Nov 1;33(11):2020-2026. doi: 10.1093/ndt/gfx364. PMID 29361078